CLINICAL TRIAL: NCT06703021
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Study of the Safety, Tolerability, and Efficacy of Increasing Optimal Doses of Aleniglipron (GSBR-1290) in Participants Living With Obesity (Body Mass Index ≥ 30 kg/m2) or Overweight (Body Mass Index ≥ 27 kg/m2) With at Least One Weight-related Comorbidity (ACCESS II)
Brief Title: A Dose-Range Study of Aleniglipron (GSBR-1290) in Participants Living With Obesity or Overweight With at Least One Weight-related Comorbidity
Acronym: ACCESS II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gasherbrum Bio, Inc., a wholly owned subsidiary of Structure Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSBR-1290-09
Record Dates: First submitted 2024-11-15; First posted 2024-11-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Overweight; Chronic Weight Management
Keywords: ACCESS II; Obesity; Overweight; GSBR-1290; Chronic weight management; Obese; Small molecule GLP-1 receptor agonist; Structure Therapeutics
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sentinel (Experimental): Participants will receive aleniglipron or placebo administered orally.
  Interventions: Drug: aleniglipron or placebo
- Cohort 1a (Experimental): Participants will receive aleniglipron or placebo administered orally.
  Interventions: Drug: aleniglipron or placebo
- Cohort 1b (Experimental): Participants will receive aleniglipron or placebo administered orally.
  Interventions: Drug: aleniglipron or placebo
- Cohort 1c (Experimental): Participants will receive aleniglipron or placebo administered orally.
  Interventions: Drug: aleniglipron or placebo

INTERVENTIONS:
Drug: aleniglipron or placebo — Drug: aleniglipron administered orally; Drug: placebo administered orally
  Arms: Cohort 1a
Drug: aleniglipron or placebo — Drug: aleniglipron administered orally; Drug: placebo administered orally
  Arms: Cohort 1b
Drug: aleniglipron or placebo — Drug: aleniglipron administered orally; Drug: placebo administered orally
  Arms: Cohort 1c
Drug: aleniglipron or placebo — Drug: aleniglipron administered orally; Drug: placebo administered orally
  Arms: Sentinel

SUMMARY:
Phase 2 clinical study will evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of various aleniglipron (GSBR-1290) dose regimens compared with placebo in participants living with obesity or overweight with ≥ 1 weight-related comorbidity, in addition to diet and exercise, over a 44-week period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* BMI ≥30 kg/m2 or BMI ≥27.0 kg/m2 and previous/current diagnosis of ≥ 1 obesity related comorbidity

Exclusion Criteria:

* Previous documented diagnosis of diabetes mellitus
* Self-reported change in body weight >5% within 3 months before Screening
* Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty, if performed >1 year prior to screening)
* Use of medications intended to promote weight loss, within 6 months prior to Screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline and week 44
Adverse events of special interest | Baseline and week 44
Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters, including hematology, plasma chemistry, coagulation, and urinalysis | Baseline and week 44
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameters: Common ECG-related variables will be assessed, including but not limited to : heart rate and QRS duration | Baseline and week 44
Number of Participants With Clinically Significant Change From Baseline in Vital Signs, including systolic and diastolic Blood Pressure, Heart Rate, Respiratory Rate, and temperature | Baseline and week 44

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to Tau (AUC0-tau) | Baseline and week 44
Maximum Observed Plasma Concentration (Cmax) of aleniglipron | Baseline and week 44
Trough Concentrations (Ctrough) of aleniglipron | Baseline and week 44
Time of Maximum Observed Plasma Concentration (Tmax) of aleniglipron | Baseline and week 44
Terminal Elimination Half-life (t1/2) for aleniglipron | Baseline and week 44

OTHER OUTCOMES:
Percent change in body weight | Baseline and week 44
Change in body weight (absolute) | Baseline and week 44
Percentage of participants who achieve ≥5% reduction in body weight at Week 44 | Baseline and week 44
Percentage of participants who achieve ≥10% reduction in body weight at Week 44 | Baseline and week 44
Percentage of participants who achieve ≥15% reduction in body weight at Week 44 | Baseline and week 44
Change in waist circumference | Baseline and week 44
Change in body mass index | Baseline and week 44
Change in patient-reported outcomes (hunger and satiety questionnaire) | Baseline and week 44
Change in HDL and LDL cholesterol | Baseline and week 44

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - ACCESS II Research Site, Glendale, California
  - ACCESS II Research Site, Montclair, California
  - ACCESS II Research Site, Valparaiso, Indiana
  - ACCESS II Research Site, West Des Moines, Iowa
  - ACCESS II Research Site, Medford, Oregon
  - ACCESS II Research Site, East Greenwich, Rhode Island
  - ACCESS II Research Site, North Charleston, South Carolina
  - ACCESS II Research Site, Dallas, Texas
  - ACCESS II Research Site, San Antonio, Texas
  - ACCESS II Research Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address a specific research question in an approved data sharing request
Supporting Information: Study Protocol
Time Frame: Data sharing requests will be considered beginning 36 months after the study publication (manuscript accepted for publication) and either 1) the product has been granted marketing authorization in at least two regulatory jurisdictions, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Researchers will submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Structure Therapeutics does not grant external requests for individual de-identified patient data for the following purposes:
  * Re-evaluating safety and efficacy end points already addressed in the product labelling,
  * Assessing safety or efficacy for an indication in current development Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a panel of external advisors. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.